CLINICAL TRIAL: NCT04519398
Title: Investigating the Involvement of ACE and Angiotensinogen Genes' Polymorphism Along With Other Thrombophilic Genotypes in Severe Forms of COVID-19 With/Without Thrombotic Events
Acronym: iGenes-COVID19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, MD, PhD, Professor, Grigore T. Popa University of Medicine and Pharmacy
Other Study IDs: GTP0051
Record Dates: First submitted 2020-08-18; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Covid19; Corona Virus Infection; Thrombosis; ARDS; Thrombophilia; Thromboses, Intracranial; Thromboses, Deep Vein; RAAS
Keywords: Covid-19; COVID-19 severity; Thrombosis; Thrombophilia; thrombophylic profile; Renin-angiotensin-aldosterone system alterations
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Thrombosis; Thrombophilia; Intracranial Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood with complete thrombophilic profile testing and RAAS components assessment through PCR (multiplex PCR and reverse hybridization of DNA to assess the presence of prothrombotic genotypes)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 patients with proved venous thrombosis: 1st group includes COVID-19 patients with proved
  * venous thrombosis (deep vein thrombosis, pulmonary embolism or venous thrombosis occurring in more atypical places such as in the veins of the brain, liver, kidney, mesenteric vein and the veins of the arms)
  * or arterial thrombosis (heart attacks, strokes)
  Interventions: Genetic: Complete thrombophilic profile testing by multiplex PCR
- Asymptomatic COVID-19 & those with mild or moderate disease: 2nd group encompasses asymptomatic patients and those with mild or moderate disease, according to current guidelines, without thrombosis: no symptoms or evidence of lower respiratory disease by clinical assessment or imaging and a SpO2 > 94%
  Interventions: Genetic: Complete thrombophilic profile testing by multiplex PCR
- Severe disease, according to Guidelines, without thrombus: 3rd group includes severe disease, according to current guidelines, without thrombosis: respiratory frequency > 30 breaths per minute, SpO2 < 94%, PaO2/FiO2 < 300 mmHg, or lung infiltrates >50%
  Interventions: Genetic: Complete thrombophilic profile testing by multiplex PCR

INTERVENTIONS:
Genetic: Complete thrombophilic profile testing by multiplex PCR — Complete thrombophilic profile testing by multiplex PCR and reverse hybridization of DNA to assess the presence of prothrombotic genotypes:
  * Factor V Leiden
  * Factor V 4070 A>G (Hr2)
  * Factor II G20210A
  * Methylenetetrahydrofolate reductase (MTHFR) C677T
  * MTHFR A1298C
  * Cystathionine β-synthase (CBS) 844ins68
  * PAI-1 4G/5G
  * Glycoprotein IIIa T1565C (HPA-1a/b)
  * ACE-DEL/INS
  * Apolipoprotein E (ApoE)
  * AGT M235T
  * Angiotensin II type 1 receptor (ATR-1) A1166C
  * Fibrinogen - 455 G>A
  * Factor XIII Val34Leu

SUMMARY:
An estimated 22% of the global population is at an increased risk of a severe form of COVID-19, while one in four coronavirus patients admitted to intensive care unit will develop a pulmonary embolism. A major public health question remains to be investigated: why COVID-19 is mild for some, critically severe for others and why only a percentage of COVID-19 patients develop thrombosis, despite the disease's proven hypercoagulable state? Patients' intrinsic characteristics might be responsible for the deep variety of disease forms.

Our study aims to assess the validity of the hypothesis according to which underlining genetic variations might be responsible for different degrees of severity and thrombotic events risks in the novel coronavirus disease.

Moreover, we suspect that prothrombotic genotypes occuring in the genes that encode angiotensin-converting enzyme (ACE-DEL/INS) and angiotensinogen (AGT M235T) are involved in the unpredictable evolution of COVID-19, both in terms of severity and thrombotic events, due to the strong interactions of SARS-CoV-2 with the renin-angiotensin-aldosterone system (RAAS). Therefore, we also aim to assess the validity of the theory according to which there is a pre-existing atypical modulation of RAAS in COVID-19 patients that develop severe forms and/or thrombosis.

Our hypothesis is based on various observations. Firstly, there is a substantial similarity with a reasonably related condition such as sepsis, for which there is a validated theory stating that thrombophilic mutations affect patients' clinical response. Secondly, racial and ethnic genetic differences are responsible for significant dissimilar thrombotic risks among various nations. Thirdly, an increase in stroke incidence has been reported in young patients with COVID-19, without essential thrombosis risk factors, favoring the idea that a genetic predisposition could contribute to increase the thrombotic and thromboembolic risk. Fourthly, the plasminogen activator inhibitor (PAI)-1 4G/5G inherited mutation was found to be responsible for a thrombotic state causing post-SARS osteonecrosis.

DETAILED DESCRIPTION:
The study's protocol will cover the following steps:

• Collected data from COVID-19 patients at admission will include:

* Descriptive general demographic data
* Previous pathologies and thrombosis risk factors
* Routine biological data (the blood routinely collected will also be used for SARS-Cov-2 specific RT-PCR exam)

Complete thrombophilic profile testing by multiplex PCR and reverse hybridization of DNA to assess the presence of prothrombotic genotypes:

* Factor V Leiden
* Factor V 4070 A G (Hr2)
* Factor II G20210A
* Methylenetetrahydrofolate reductase (MTHFR) C677T
* MTHFR A1298C
* Cystathionine β-synthase (CBS) 844ins68
* PAI-1 4G/5G
* Glycoprotein IIIa T1565C (HPA-1a/b)
* ACE-DEL/INS
* Apolipoprotein E (ApoE)
* AGT M235T
* Angiotensin II type 1 receptor (ATR-1) A1166C
* Fibrinogen - 455 G A
* Factor XIII Val34Leu SpO2, respiratory rate, PaO2/FiO2 RAAS components

  * Imagistic procedures (chest X-ray or CT)

    * All patients with a positive SARS-CoV-2 PCR test will be included
    * Patients will be divided into three groups depending on disease severity and the presence of thrombotic state:
  * 1st group includes COVID-19 patients with proved
* venous thrombosis (deep vein thrombosis, pulmonary embolism or venous thrombosis occurring in more atypical places such as in the veins of the brain, liver, kidney, mesenteric vein and the veins of the arms)
* or arterial thrombosis (heart attacks, strokes)

  * 2nd group encompasses asymptomatic patients and those with mild or moderate disease, according to current guidelines, without thrombosis: no symptoms or evidence of lower respiratory disease by clinical assessment or imaging and a SpO2 ≥ 94%
  * 3rd group includes severe disease, according to current guidelines, without thrombosis: respiratory frequency > 30 breaths per minute, SpO2 < 94%, PaO2/FiO2 < 300 mmHg, or lung infiltrates >50%

    * Statistical methods will be employed to check for significant differences between prothrombotic mutations frequency and RAAS components levels for the three groups

ELIGIBILITY:
Inclusion Criteria:

* All hospitalized patients with cough, fever, myalgia - with confirmed COVID-19 infection • All patients with a positive SARS-CoV-2 PCR test

Exclusion Criteria:

* Patient refusal
* Uncertain tests results
* Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with COVID-19 and thrmbotic events or, Patients with COVID-19 & no thrombotic events but with a severe form Patients with COVID-19 & no thrombotic events and no or mild symptoms
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-02-17 (Estimated); Study Completion 2021-08-18 (Estimated)

PRIMARY OUTCOMES:
Number of patients with thrombophilic profile alterations | One year
  The difference of prothrombotic genotypes frequency between the three groups

SECONDARY OUTCOMES:
Number of patients with RAAS components alterations | One year
  The differences of RAAS components levels between the three groups

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Professor, Study Chair — Gr T Popa University of Medicine and Pharmacy Iasi ROMANIA
Locations (1):
- University of Medicine and Pharmacy Gr T. Popa Iasi, Romania, Iași, Romania

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR